CLINICAL TRIAL: NCT05656859
Title: Prevalence of Eating Disorder Symptomatology Among Outpatients Referred to Health Promotion from Somatic Hospital Departments
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Tobias Christensen, Principal Investigator, Aalborg University Hospital
Other Study IDs: F2022-088
Record Dates: First submitted 2022-12-06; First posted 2022-12-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Population Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Descriptive study
  Interventions: Behavioral: Single group

INTERVENTIONS:
Behavioral: Single group — Survey

SUMMARY:
The Department of Health Promotion at Aalborg University Hospital gets patients referred from all the hospital's departments. The Department of Health Promotion offers lifestyle courses to aid preventing disease relapses and further comorbidities to patients referred to other ambulatory treatments at the hospital. For most patients this also includes weight loss, but the primary goal is lifestyle change regarding eating and exercise habits to improve overall health state. Since it is known that eating disorders commonly occurs in individuals seeking help for weight loss, and that the prevalence is larger than in the background population, we also suspect that eating disorders would commonly occur among patients referred to the Department of Health Promotion. Therefore, we aim to investigate the prevalence of eating disorders among patients referred to lifestyle courses at the Department of Health Promotion.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the Department of Health Promotion at Aalborg University Hospital, Denmark

Exclusion Criteria:

* Under age 18
* Not able to read and understand Danish
* Not able to recieve mail in the danish digital postbox, e-Boks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the Department of Health Promotion
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination Questionnaire (EDE-Q) | 10 minutes
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-reported questionnaire adapted from the semi-structured interview Eating Disorder Examination (EDE) and designed to assess the range and severity of features associated with a diagnosis of eating disorder using 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and a global score.
  The EDE-Q generates two types of data: frequency data on key behavioural features of eating disorders in terms of number of episodes of the behaviour, and subscale scores reflecting the severity of characteristics of eating disorders.
  Higher scores on the global scale and subscales denote more problematic eating behaviours and attitudes.

SECONDARY OUTCOMES:
Binge Eating Disorder Questionnaire (BED-Q) | 5 minutes
  The Binge Eating Disorder Questionnaire (BED-Q) is a 9-item self-reported questionnaire. Items are rated on a 5-point Likert-type rating scale. Scores range between 0-32 and higher scores denote more problematic binge eating disorder. A diagnostic score that determine patient is diagnosed with Binge Eating Disorder or not can be calculated. 1 item rated "yes" or "no and other items are used to calculated a diagnostic score.
Grazing Questionnaire (GQ) | 5 minutes
  Grazing Questionnaire (GQ) is a 8-item self-reported questionnaire to measure behaviours and cognitions specific to grazing. Items are rated on a 5-point Likert-type rating scale where higher scores represent more grazing behaviours and cognitions. Scores are summes to form a total score (range: 0-32).

OTHER OUTCOMES:
The 5-level EQ-5D version (EQ-5D-5L) | 5 minutes
  Self-reported quality of life questionnaire. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University Hospital, Aalborg, North of Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No